CLINICAL TRIAL: NCT01438918
Title: A Long-term, Confirmatory, Phase 3, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study To Investigate The Safety And Efficacy Of Orally Administered Sd-6010 In Subjects With Symptomatic Osteoarthritis Of The Knee
Brief Title: X-Ray Study Investigating The Safety And Efficacy Of SD-6010 In Subjects With Osteoarthritis Of The Knee
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6171017
Record Dates: First submitted 2011-09-13; First posted 2011-09-22 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; X-ray; Joint Space Narrowing
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — cindunistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 mg (Active Comparator): High dose active comparator
  Interventions: Drug: SD-6010
- 50 mg (Active Comparator): Low dose active comparator
  Interventions: Drug: SD-6010
- Placebo (Placebo Comparator): Placebo comparator to be used for control purposes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SD-6010 — 200 mg tablets once a day for 2 years
  Arms: 200 mg
Drug: SD-6010 — 50 mg tablets once a day for 2 years
  Arms: 50 mg
Drug: Placebo — Placebo tablets once a day for 2 years
  Arms: Placebo

SUMMARY:
The objective of this 2-year study is to evaluate the safety, tolerability and disease modifying efficacy of SD 6010, an inhibitor of inducible nitric oxide synthase (iNOS). The efficacy of SD-6010 will be evaluated by radiography using joint space narrowing in the medial tibiofemoral compartment of the study knee as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged >= 40 years Diagnosed with knee OA (ACR definition of OA) Radiographic evidence of OA in the study knee

Exclusion Criteria:

A diagnosis of any other rheumatic disease Current conditions in the study knee that would confound efficacy Selected, traditional clinical safety and laboratory parameters

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To assess the progression rate of joint space narrowing in the study knee of subjects with knee OA over a 24-month period | 24 months

SECONDARY OUTCOMES:
Clinical benefit of SD 6010 will be measured from changes in response from baseline to 24 months in 7 patient reported outcomes (PRO), including, but not limited to, WOMAC, pain VAS, ICOAP, KOOS. | 24 months
Total analgesic medication burden for OA in the study knee will be compared back to baseline of an increased, sustained use of standard background and/or rescue medication for more than 30 days as measured at the Month 12 and 24 visits | 24 months
Safety: Change from baseline to M24 in vital signs (blood pressure, heart rate) measurements will be assessed | 24 months
Safety: Change from baseline to M24 in ECG abnormalities | 24 months
Safety: In a subset of subjects: Change from baseline on average as assessed by 24-h ambulatory blood pressure monitoring (ABPM) at months 3 and 6 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6171017&StudyName=X-Ray%20Study%20Investigating%20The%20Safety%20And%20Efficacy%20Of%20SD-6010%20In%20Subjects%20With%20Osteoarthritis%20Of%20The%20Knee